CLINICAL TRIAL: NCT06050265
Title: Glucose Evaluation Through Continuous Glucose Monitors in Polycystic Ovary Syndrome
Acronym: GEMS-PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-39852
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries; Dysglycemia; Insulin Resistance
Keywords: continuous glucose monitor
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention arm - CGM (Experimental): Participants randomized to intervention arm will be given standard of care nutrition and exercise counseling to optimize weight, nutrition and glycemic status AND will be asked to wear a DEXCOM CGM for 90 days.
  Interventions: Device: DEXCOM Continuous Glucose Monitor (CGM)
- Control arm (No Intervention): Participants randomized to control arm will ONLY be given standard of care nutrition and exercise counseling to optimize weight, nutrition and glycemic status.

INTERVENTIONS:
Device: DEXCOM Continuous Glucose Monitor (CGM) — Dexcom CGMs are placed every 10 days and provide a continuous assessment of blood glucose.
  Arms: Intervention arm - CGM

SUMMARY:
PCOS is the most common endocrine disorder of reproductive aged women. In addition to menstrual and endocrine abnormalities, PCOS is characterized by insulin resistance and glycemic dysregulation. The pattern of glycemic abnormalities among patients with PCOS may be different than the general population, as evidenced by invasive, time consuming, and costly procedures such as the euglycemic clamp or oral glucose tolerance test. Continuous glucose monitoring (CGM) offers an opportunity to evaluate glycemic status in real world conditions. Furthermore, use of a CGM has been found to improve glycemic status among those with prediabetes and diabetes, but little is known about utility among patients with PCOS. The investigators thus seek to 1) characterize glycemic status using CGM among patients with PCOS and 2) assess the impact of CGM use on metabolic and reproductive health in patients with PCOS.

DETAILED DESCRIPTION:
Study synopsis:

Recruitment:

* PCOS participants will be recruited from those who are being seen or have previously been seen at the UCSF multidisciplinary PCOS clinic.
* Non-PCOS participants will be recruited from patients being seen at the UCSF Center for Reproductive Health for other clinical evaluations or research projects.

Study protocol:

Aim 1:

Pre-DEXCOM evaluation:

PCOS participants:

* As part of routine clinical care all PCOS participants will have had the following procedures completed:
* Blood work for fasting and 2 hour glucose/insulin, hgba1c, CRP, lipid panel, liver enzymes, SHBG, free and total testosterone, DHEAS, androstenedione, 17-OH-Progesterone, prolactin, TSH, FSH, LH, E2, estrone, Vit D.
* Screening questionnaires on physical exercise using validated International Physical Activity Questionnaire
* In person clinical evaluation including physical exam and history.
* In person transvaginal ultrasound assessment.
* The above are part of standard of care screening for patients with concern for PCOS and are currently routinely completed at the UCSF Center for Reproductive Health in this setting.
* Participants will also be asked to complete a 10 question validated fatigue assessment scale (FAS)

Non-PCOS participants:

* Participants will have blood work for fasting and 2 hour glucose/insulin, hgba1c, CRP, lipid panel, liver enzymes, SHBG, free and total testosterone, DHEAS, androstenedione, 17-OH- Progesterone, prolactin, TSH, FSH, LH, E2, estrone, Vit D obtained.
* Screening questionnaires on physical exercise using validated International Physical Activity Questionnaire will be obtained.
* Participants will be asked to complete the same intake questionnaires that PCOS participants complete as part of standard of care practices in the UCSF multidisciplinary PCOS clinic, which include questions on ethnicity, family, medical, and social history.
* If blood work was not completed as part of standard of care for routine clinical evaluation or as part of a previously completed research study in which the patient provided consent for their data to be used in other trials, the above labs will be collected and paid for by the research protocol.
* Participants will also be asked to complete a 10 question validated fatigue assessment scale (FAS)

Procedures:

DEXCOM evaluation:

* PCOS and non-PCOS participants will be given a DEXCOM CGM to wear for 10 days. During this time they will be blinded to the results of the DEXCOM.
* Participants will be asked to complete the automated self-administered 24-hour dietary assessment (ASA24) tool, which is a web based, validated 24 hour dietary record program, produced by the National Cancer Institute (NCI)/Nation Institute of Health and made available free of charge to researchers.
* As part of the ASA24 participants will also be asked about their sleep quality the night prior to their dietary record. See attached module.
* All participants will be asked to complete the ASA24 during a 24 hour period while wearing the CGM.

Aim 2:

Recruitment:

* From those participants with PCOS recruited for Aim 1, a subgroup with evidence of dysglycemia (as outlined in the inclusion criteria) will be recruited for aim 2.
* Participants will be randomized in a 3:1 fashion to intervention with CGM vs control.

Procedures:

Intervention group:

* All participants will receive standard of care nutrition and exercise advice from a trained registered dietician.
* Participants randomized to the intervention arm will also receive education on how to use and monitor blood glucose using the DEXCOM G7 CGM and associated phone application.
* Participants will be asked to use a CGM continuously for 90 days.
* After 90 days blood work for fasting and 2 hour glucose/insulin, hgba1c, CRP, lipid panel, liver enzymes, SHBG, free and total testosterone, DHEAS, androstenedione, 17-OH-Progesterone, prolactin, TSH, FSH, LH, E2, estrone, Vit D will be obtained.
* After 90 days participants will also be asked to repeat a 10 question validated fatigue assessment scale (FAS)
* After 90 days participants will be asked about their menstrual cycle pattern over the 90 day period

Control group:

* All participants will receive standard of care nutrition and exercise advice from a trained registered dietician.
* After 90 days blood work for fasting and 2 hour glucose/insulin, hgba1c, CRP, lipid panel, liver enzymes, SHBG, free and total testosterone, DHEAS, androstenedione, 17-OH-Progesterone, prolactin, TSH, FSH, LH, E2, estrone, Vit D will be obtained.
* After 90 days, participants in the control group will be given the opportunity to receive CGM devices to monitor blood glucose up to 30 days with education on how to use the device and associated phone application to monitor blood glucose.
* After 90 days participants will also be asked to repeat a 10 question validated fatigue assessment scale (FAS)
* After 90 days participants will be asked about their menstrual cycle pattern over the 90 day period

Data Management:

Clinical and laboratory data will be stored in a Research Electronic Data Capture (REDCap) system designed by Dr. Huddleston and research staff. Fields will be designed by study coordinators with input from key investigators. Our team has extensive experience with REDCap architecture and utilization.

ELIGIBILITY:
Inclusion Criteria:

For aim 1:

* Aged 18-45
* Female sex
* Agree to wear a CGM for 10 days
* Have access to an apple or android smart phone for CGM monitoring
* Are able to be characterized as PCOS or non-PCOS using the 2003 Rotterdam criteria for PCOS of 2 or more of the following: 1) biochemical or clinical hyperandrogenism, 2) polycystic ovarian morphology on transvaginal ultrasound, and/or 3) oligo-amenorrhea

For aim 2:

* All of the inclusion criteria for aim 1
* Meet 2003 Rotterdam criteria for PCOS as above
* Evidence of baseline glycemic dysregulation including any of the following: 1) elevated fasting glucose (100-125 mg/dL), 2) elevated 2 hour glucose (140-200 mg/dL), 3) elevated fasting insulin (>10 mIU/mL), 4) elevated 2 hour insulin (>40 mIU/mL), 5) elevated Hgba1c (5.7- 6.4)

Exclusion Criteria:

For both aims 1 and 2:

* Use of metformin or other anti-diabetic agents
* Diagnosis of type I or II diabetes mellitus (including those found to have fasting glucose >126, 2 hour glucose >200, Hgba1c >6.5)
* Prior or current use of CGM

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-11-29 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Difference between change in hemoglobin A1C | 90 days
  Difference between change in hemoglobin A1C for 2 treatment arms from baseline to after 90 days

SECONDARY OUTCOMES:
Difference between change in fasting insulin | 90 days
  Difference between change in fasting insulin for 2 treatment arms from baseline to after 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Heather G Huddleston, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Center for Reproductive Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tatulashvili S, Baptiste Julla J, Sritharan N, Rezgani I, Levy V, Bihan H, Riveline JP, Cosson E. Ambulatory Glucose Profile According to Different Phases of the Menstrual Cycle in Women Living With Type 1 Diabetes. J Clin Endocrinol Metab. 2022 Sep 28;107(10):2793-2800. doi: 10.1210/clinem/dgac443. PMID 35869507
- [Background] Legro RS, Castracane VD, Kauffman RP. Detecting insulin resistance in polycystic ovary syndrome: purposes and pitfalls. Obstet Gynecol Surv. 2004 Feb;59(2):141-54. doi: 10.1097/01.OGX.0000109523.25076.E2. PMID 14752302
- [Background] Diamanti-Kandarakis E, Dunaif A. Insulin resistance and the polycystic ovary syndrome revisited: an update on mechanisms and implications. Endocr Rev. 2012 Dec;33(6):981-1030. doi: 10.1210/er.2011-1034. Epub 2012 Oct 12. PMID 23065822